CLINICAL TRIAL: NCT07319364
Title: An Observational, Real-World Study Evaluating Fecal Microbiota Transplantation for the Prevention/Reduction of Chemotherapy/Targeted Therapy-Induced Gastrointestinal Symptoms in Patients With Gastrointestinal Cancers.
Brief Title: A Real-World Study of Fecal Transplants for Cancer Therapy Side Effects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1390
Record Dates: First submitted 2025-11-17; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Fecal Microbiota Transplantation (FMT); Gastrointestinal Neoplasms; Antineoplastic Agents; Drug-related Side Effects and Adverse Reactions
Keywords: Fecal Microbiota Transplantation; Gastrointestinal Neoplasms; Antineoplastic Agents; Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Gastrointestinal Neoplasms; Drug-Related Side Effects and Adverse Reactions | interventions — Fecal Microbiota Transplantation; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in the control group continued their original chemotherapy/targeted therapy regimen, with each treatment cycle lasting 3 weeks, for a total of 5 cycles. Treatment efficacy was assessed after every 2 cycles.
- Experimental Group (Experimental): Patients in the FMT group received treatment starting from the fourth cycle on top of their existing regimen. They underwent one FMT treatment within 3 days prior to chemotherapy/targeted therapy during the fourth, sixth, and eighth cycles (weeks 3, 9, and 15 after study initiation). Each transplant consisted of approximately 40g of donor gut microbiota encapsulated in capsules. The capsules were administered orally, typically at a dose of 2-3 capsules (1g/capsule) every 3-5 minutes, totaling 40 capsules per dose for a total of 120 capsules. Treatment cycles were conducted every 3 weeks, with therapeutic efficacy assessed after every 2 cycles.
  Interventions: Biological: Fecal microbiota transplantation (FMT)

INTERVENTIONS:
Biological: Fecal microbiota transplantation (FMT) — Building upon the existing treatment regimen, starting from the fourth cycle, one FMT treatment was administered within 3 days prior to chemotherapy/targeted therapy during the fourth, sixth, and eighth cycles (weeks 3, 9, and 15 after study initiation). Each transplant consisted of approximately 40g of donor intestinal bacteria encapsulated in capsules. The capsules were administered orally, typically at a dose of 2-3 capsules (1g/capsule) every 3-5 minutes, totaling 40 capsules per dose for a total of 120 capsules. Treatment cycles were conducted every 3 weeks, with therapeutic efficacy assessed after every 2 cycles.
  Other Names: Chemotherapy; Targeted Therapy
  Arms: Experimental Group

SUMMARY:
The goal of this clinical trial is to learn if fecal microbiota transplantation can treat in Gastrointestinal cancer patients with chemotherapy / targeted gastrointestinal symptoms. The main question it aims to answer is: To evaluate the effect of fecal microbiota transplantation (FMT) on gastrointestinal tract in patients with gastrointestinal tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, gender not restricted;
2. Estimated survival time ≥ 3 months;
3. Confirmed diagnosis of gastrointestinal tumors by pathological examination, including esophageal cancer, gastric cancer, colon cancer, rectal cancer, etc.;
4. TNM staging of cancer in patients is Stage IV;
5. Having undergone PD-1 or PD-L1 testing;
6. Planned to receive the 4th cycle of chemotherapy/targeted therapy;
7. Occurrence of gastrointestinal adverse reactions (including but not limited to diarrhea, constipation, vomiting, nausea, etc.) within 3 cycles of conventional chemotherapy/targeted therapy;
8. Patients are able and willing to sign the informed consent form and complete follow-up;
9. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 1-3;
10. Use of oral/intravenous broad-spectrum antibiotics with caution within 3 days;
11. Patients are able to swallow capsules without chewing;
12. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 1-3;
13. Laboratory test results during the screening period indicate that the subjects have sufficient organ function.

Exclusion Criteria:

1. Patients with major organ dysfunction or even failure, including but not limited to cardiac insufficiency or heart failure, renal insufficiency or renal failure, and hepatic insufficiency/hepatic failure;
2. Uncontrolled or severe infections;
3. Known history of psychotropic substance abuse, alcoholism, and drug abuse;
4. Patients with severe infections complicated with septicemia or sepsis;
5. Patients with a history of severe allergic reactions or a known allergy to the components of liquid live bacteria enteric-coated capsules;
6. Patients with active viral infections;
7. Female subjects with a positive pregnancy test, lactating female subjects, and women of childbearing age who refuse to use contraceptive measures during the entire observation period (15 weeks);
8. Patients with gastrointestinal perforation and/or fistula;
9. Other conditions deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and improvement rate of chemotherapy/targeted therapy-induced gastrointestinal symptoms in patients with gastrointestinal cancers | At 8 weeks post-FMT
  This outcome measure assesses the incidence (grade ≥1 per CTCAE 5.0) and improvement rate (≥1-grade reduction in symptom severity or ≥30% decrease in EORTC QLQ-C30 scores) of chemotherapy/targeted therapy-induced gastrointestinal (GI) symptoms (e.g., nausea, vomiting, diarrhea) in patients with gastrointestinal cancers receiving fecal microbiota transplantation (FMT), as determined by scale scores and adverse event grading at baseline and post-treatment follow-up.

SECONDARY OUTCOMES:
The incidence and improvement rate of gastrointestinal (GI) symptoms in patients with gastrointestinal cancers | At 4 weeks post-FMT
  This outcome measure assesses the incidence (grade ≥1 or exacerbation of baseline symptoms per CTCAE 5.0) and improvement rate (≥1-grade reduction in symptom severity or ≥30% decrease in GSRS scores) of chemotherapy/targeted therapy-induced gastrointestinal symptoms (e.g., nausea, vomiting) in patients with gastrointestinal cancers receiving FMT.
Changes in Gut Microbiota Diversity Indices | At 4, 8 weeks post-FMT
  This secondary outcome measure assesses changes in gut microbiota α-diversity (Shannon Index and Simpson Index, dimensionless, reflecting microbial richness and evenness) and β-diversity (Bray-Curtis dissimilarity and Jaccard distance, dimensionless, reflecting differences in community structure) after the 4th and 8th cycles of fecal microbiota transplantation (FMT) combined with chemotherapy/targeted therapy in patients with gastrointestinal cancers, using 16S rDNA high-throughput sequencing (V3-V4 region, Illumina NovaSeq platform) to evaluate FMT's regulatory effect on gut microbiota diversity during anti-tumor treatment.
Correlation Between Changes in Gut Microbiota Abundance and Improvement of Gastrointestinal Symptoms | At 8 weeks post-FMT
  This secondary outcome measure explores the correlation between dynamic changes in gut microbiota abundance (relative abundance % at phylum/genus/species levels; absolute abundance of key taxa, copies/μg fecal DNA, detected via 16S rDNA sequencing and qPCR) at baseline, 4th and 8th treatment cycles, and improvement of chemotherapy/targeted therapy-induced GI symptoms (≥30% GSRS score reduction or ≥1-grade CTCAE relief) in gastrointestinal cancer patients receiving FMT + anti-tumor treatment, using Spearman/Pearson coefficients and subgroup analyses by symptom type to reveal the underlying mechanism.

OTHER OUTCOMES:
Comparison of Changes in Serum Tumor Markers, IL-6, IL-8, Soluble Tumor Necrosis Factor Receptor 1 (sTNFR1), CRP, and Neutrophil (NE) Ratio Before and After FMT Combined with Chemotherapy/Targeted Therapy | At 8 weeks post-FMT
  This secondary outcome measure compares changes in serum tumor markers (e.g., CEA, CA19-9), inflammatory factors (IL-6, IL-8, soluble Tumor Necrosis Factor Receptor 1 [sTNFR1], CRP), and Neutrophil (NE) Ratio before and after fecal microbiota transplantation (FMT) combined with chemotherapy/targeted therapy in gastrointestinal cancer patients, by detecting serum samples to evaluate the treatment's impact on tumor burden and systemic inflammatory status.
Comparison of Changes in Blood Lymphocyte Subsets (e.g., B Cells, NK Cells, Monocytes) Before and After FMT Combined with Chemotherapy/Targeted Therapy | At 8 weeks post-FMT
  This outcome measure compares changes in the count and proportion of lymphocyte subsets (e.g., B cells, NK cells, monocytes) by detecting blood samples from gastrointestinal cancer patients before and after fecal microbiota transplantation (FMT) combined with chemotherapy/targeted therapy, to evaluate the treatment's regulatory effect on patients' immune function.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Zhejiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No